CLINICAL TRIAL: NCT04365855
Title: The Olmsted NAFLD Epidemiology Study (TONES)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alina M. Allen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-004848
Record Dates: First submitted 2020-04-09; First posted 2020-04-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Elasticity Imaging Techniques; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: We will invite adult Olmsted County residents with research authorization, identified based on a random search of the Rochester Epidemiology Project database. We plan to accrue 800 participants. Based on literature estimates, approximately 25-30% of adults will be at risk for NAFLD due to overweight/obese status. Participants will undergo tests for NAFLD screening: blood tests, Magnetic Resonance Imaging/Elastography and electrocardiogram. Those identified with fatty liver will undergo Transient elastography and liver biopsy for disease severity assessment. These results will be used to validate a machine learning model of NAFLD diagnosis and liver disease severity which uses the participants clinical and laboratory data (noninvasive electronic health records). The cohort will be followed for 5 years, when they will return for repeat imaging and blood tests to monitor for incident NAFLD, liver disease progression and outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects at risk for NAFLD (Other): Adult Olmsted County residents identified as at risk for NAFLD will receive Magnetic Resonance Imaging (MRE,) blood tests,and possible biopsy.
  Interventions: Diagnostic Test: Magnetic Resonance Elastography; Other: Blood draw; Procedure: Liver biopsy; Procedure: Fibro Scan

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography — Combines MRI imaging with sound waves to create a visual map (elastogram) showing the stiffness of body tissues.
Other: Blood draw — Clinical blood tests with a focus on liver function parameters and diabetes
Procedure: Liver biopsy — If indicated per MRE results a biopsy will be taken of the liver.
Procedure: Fibro Scan — If indicated per MRE results a fibroscan will be performed of the liver.

SUMMARY:
Researchers are assessing the prevalence of Non-alcoholic Fatty Liver Disease (NAFLD) and Nonalcoholic Steatohepatitis (NASH) in the population and assembling a well-characterized cohort of adults with NAFLD and NASH to validate models of NAFLD diagnosis and determine long-term outcomes.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is the most common cause of chronic liver disease in the world and a major public health issue in the US. Recent information on the prevalence of NAFLD in general and Non-Alcoholic Steatohepatitis (NASH) with fibrosis in particular is very scarce. Such information is crucial for defining the epidemiology of NAFLD, identifying risk factors for advanced fibrosis and longitudinal outcomes. This study will enroll a random sample of adults from Olmsted County, Minnesota, to validate machine learning models for NAFLD diagnosis and disease severity. These data would be fundamental for the development of screening strategies in the community, which are urgently needed for early diagnosis of liver fibrosis and therapeutic interventions before cirrhosis develops.

ELIGIBILITY:
Inclusion Criteria:

* Olmsted County residents at the time of search
* Age 18 or older
* No personal history of NAFLD diagnosis (administrative codes)

Exclusion Criteria:

* Alcohol in excess (more than 20 gm per week in women and 30 gm per week in men)
* Currently pregnant
* Have contraindications to MRI (MRI incompatible implanted devices, severe claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD and NASH in the population | 5 years
  Number of subjects with NAFLD and NASH determined by the MRE

SECONDARY OUTCOMES:
Long-term health outcomes | 5 years
  Number of participants to experience the development of NAFLD, NASH, NASH cirrhosis complications, liver transplant, cardiovascular events, cancers or death

CONTACTS AND LOCATIONS:
Overall Officials: ALINA M ALLEN, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials